CLINICAL TRIAL: NCT01539551
Title: Investigation of the Role of Brain Natriuretic Peptide and Lactate in Early Goal-directed Therapy for Patients With Severe Sepsis and Septic Shock
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201111015RIB
Record Dates: First submitted 2012-02-21; First posted 2012-02-27 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-03

CONDITIONS: Sepsis; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Lactic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood(serum/plasma)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: sepsis and septic shock patients
  Interventions: Other: check BNP and lactate

INTERVENTIONS:
Other: check BNP and lactate — we will collect patients's blood samples on Day 0, Day1 and Day2

SUMMARY:
B-type natriuretic peptide (BNP) is a cardiac neurohormone which rapidly released by the ventricle in response to myocardial stretch. BNP has been used as a biomarker of sepsis related cardiac dysfunction and volume overload in critical ill patients. It is also a marker associated with prognosis in patients with severe sepsis and septic shock. However, the clinical utility of BNP level in management of early severe sepsis and septic shock over the first 48 hours is not clear. Besides, Lactate represents as a maker of tissue hypoperfusion, which has been used as a guide therapy for sepsis patients and high serum lactate level is independently associated with mortality in severe sepsis. Today, in management of early severe sepsis and septic shock, current guideline emphasize the early goal-directed therapy (EGDT) with achieving the central venous pressure (CVP) level 8-12 mmHg by fluid support first, then targeting the next goal to maintain mean airway pressure (MAP) at least 65 mmHg by vasopressor agent (ie, Norepinephrine) and finally keeping central venous oxyhemoglobin saturation (ScvO2) > 70% via optimal Hct > 30% and dobutamine usage within first 6 hours of emergency department admission. However, the role of BNP and lactate in patients with severe sepsis and septic shock with or without myocardial dysfunction under EGDT management are not clear.

The investigators will conduct a prospective observational study to investigate the change of BNP and Lactate within 48 hours in early severe sepsis and septic shock under EGDT management, their association of cardiac dysfunction and their role in predicting various clinical outcome. The investigators also want to see if BNP and lactate could be useful tools to guide the adjustment of optimal fluid supply and the timing of inotropic agent intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old
* Severe sepsis with or without septic shock

Exclusion Criteria:

1. Previous known heart failure or cardiomyopathy history
2. Acute coronary syndrome
3. Clinical pulmonary hypertension with various cause (iPAH, congenital heart disease, CTEPH, COPD with cor pulmonale)
4. Patients with acute pulmonary embolism
5. Chronic Af with LVH
6. Acute cerebral vascular event
7. Respiratory failure with high PEEP > 10 cmH2O)
8. Various cancer with distant metastasis
9. Patients with Bosmin therapy
10. Patients received CPR (IHCA or OHCA)
11. Massive GI bleeding or hypovolemic shock
12. Pregnancy
13. Contraindication to central venous catheterization
14. Drug overdose
15. Burn injury, trauma patients
16. A requirement for immediate surgery
17. Liver cirrhosis child C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe sepsis with or without septic shock
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | 6 months
  ICU mortality, hospital mortality,

SECONDARY OUTCOMES:
Morbidity | 6 months
  AKI RIFLE stage, evidence of UGI bleeding,Ventilator days,Length of ICU stay,

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Fu Chen, MD, Principal Investigator — National Taiwan University Hospital Yulin- branch
Locations (1):
- National Taiwan University Hospital Yulin Branch, Yulin, Taiwan, Taiwan